CLINICAL TRIAL: NCT05697692
Title: An Investigation of Clinical Outcomes and Inflammatory Response to Heparin Free Extracorporeal Membrane Oxygenation Support During Clinical Lung Transplantation - a Prospective Double-blind Randomised Feasibility Study
Brief Title: Heparin-free Extracorporeal Membrane Oxygenation Support During Clinical Lung Transplantation
Acronym: zero-hep
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Schwarz, PI, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2128/2021
Record Dates: First submitted 2023-01-12; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Lung Transplantation
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Saline 0.9%
  Interventions: Drug: Placebo
- Heparin sodium (Active Comparator): 70 international units (IU)/kg Heparin sodium
  Interventions: Drug: Heparin sodium

INTERVENTIONS:
Drug: Heparin sodium — Lung transplantation on central veno-arterial ECMO with standard additional heparin
  Arms: Heparin sodium
Drug: Placebo — Lung transplantation on central veno-arterial ECMO without additional heparin
  Arms: Placebo

SUMMARY:
The aim of this investigation is to compare two different anti-coagulation strategies in clinical lung transplantation where lung implantations are all routinely done on veno-arterial (VA) extracorporeal membrane oxygenation (ECMO) support at the investigators' institution. No heparinization (Zero-Hep) will be compared to standard low-dose heparinization (Standard). Traditionally, the Vienna group has used a standard low-dose heparin protocol with unfractionated heparin (UFH) administered as a bolus upon ECMO cannulation. With heparin-coated tubing and intraoperative ECMO flow never falling below 1 L/min, the likelihood of thromboembolic events is believed to be negligible. To date, the investigators have not experienced any thromboembolic events during intra-operative ECMO use. On the other hand, the use of UFH entails an increased risk for bleeding, so it follows that avoidance of additional heparin may be beneficial. Generally, risks and benefits of heparinization during these short procedures have not yet been thoroughly analyzed. This study will investigate the feasibility of running heparin free VA-ECMO support during clinical lung transplantation and its effect on clinical outcomes and inflammatory response comparing 40 patients receiving a standard dose of heparin versus 40 patients receiving placebo in a randomized, double-blind study design.

ELIGIBILITY:
Inclusion Criteria:

* Double lung transplantation
* Age of 18 or older at the time of the procedure

Exclusion Criteria:

* Single lung transplantation
* Re-transplantation
* Previous major thoracic surgery (excluding pleural drainage, video-assisted thoracoscopic - (VATS) biopsy)
* ECMO bridge to transplantation
* Coronavirus(COVID) - acute respiratory distress syndrome (ARDS) as transplant indication
* Pre-operative anti-coagulation/anti-platelet treatment
* Paediatric transplantation
* Multi-organ transplantation
* Active pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Arterial thromboembolic events | From time of intraoperative ECMO initiation, assessed uo to 3 weeks post-transplant
  Including myocardial infarction, mesenteric infarction, hepatic infarction, spleen infarction, limb ischemia, cerebral stroke including transient ischemic attack
Venous thromboembolic events | From time of intraoperative ECMO initiation, assessed up to 3 weeks post-transplant
  deep vein thrombosis, pulmonary embolism, cerebral venous or cavernous sinus thrombosis
Circuit-related thrombosis | From time of intraoperative ECMO initiation assessed until intraoperative ECMO decannulation
  requiring ECMO oxygenator exchange

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Hoetzenecker, MD PhD, Principal Investigator — Medical University of Vienna - Dept. of Thoracic Surgery
Locations (1):
- Medical University of Vienna - Dept. of Thoracic Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No